CLINICAL TRIAL: NCT07085559
Title: Safety and Efficacy of Metabolically Armed BCMA CAR-T Cells (Meta10-BCMA) in the Treatment of r/r Plasma Cell Neoplasms Clinical Research
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM-META10-BCMA-11
Record Dates: First submitted 2025-07-14; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma (MM); Plasma Cell Leukemia (PCL); AL Amyloidosis (AL)
Keywords: Meta10-BCMA; CAR-T Cells Therapy; r/r plasma cell neoplasms
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Metabolically Armed BCMA CAR-T cells. (Experimental): Patients undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CAR-T cells infusion.
  The study will design metabolically armed BCMA CAR-T cells(Meta10-BCMA) with different structures. A dose of Meta10-BCMA CAR-T cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed BCMA CAR-T cells.

INTERVENTIONS:
Drug: Metabolically Armed BCMA CAR-T cells. — Each subject receive metabolically armed BCMA CAR- T cells by intravenous infusion.
  Other Names: Meta10-BCMA

SUMMARY:
A Study of Metabolically Armed BCMA CAR-T Cells Therapy for Patients With Relapsed and/or Refractory Plasma Cell Neoplasms.

DETAILED DESCRIPTION:
This is an open-label study. This study is indicated for relapsed or refractory Plasma Cell Neoplasms.The selections of dose levels and the number of subjects are based on clinical trials of similar products and the outcomes of our preliminary clinical studies.

1. Main research objectives:

   To evaluate the safety and tolerability of metabolically armed BCMA CAR-T Cells in the treatment of r/r plasma cell neoplasms.
2. Secondary research objectives:

(1)To evaluate the pharmacokinetic (PK) and pharmacodynamics (PD) characteristics of metabolically armed BCMA CAR-T cells after infusion.

(2) To evaluate tumor remission after infusion of metabolically armed BCMA CAR-T Cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 75 years old, male or female. The subject or his/her guardian voluntarily signed the informed consent;
* Subjects with relapsed or refractory Plasma Cell Neoplasms（including Multiple Myeloma, Plasma Cell Leukemia, AL Amyloidosis）according to IMWG criteria and have had at least 3 prior lines of therapy (including chemotherapy based on proteasome inhibitors and immunomodulatory agents). Disease progression must be documented during or within 12 months following the most recent anti-myeloma treatment (for subject whose last-line treatment was CAR-T, disease progression was not limited to occurring within 12 months after treatment).
* Evidence of cell membrane BCMA expression, as determined by a validated immunohistochemistry (IHC) or flow cytometry of tumor tissue.
* The subjects were unable to receive autologous hematopoietic stem cell transplantation treatment, or relapsed after autologous hematopoietic stem cell transplantation, and the researchers determined that treatment was needed.
* ECOG performance score 0-2 (except for subjects with central nervous system invasion, which needs to be confirmed by the investigator).
* Estimated life expectancy≥12 weeks.
* Subjects should have adequate organ function:

  1. Complete blood count (CBC) test [the following criteria should be met within 24 hours prior to apheresis, and supportive treatment such as transfusion, platelet transfusion, cell growth factor (except recombinant erythropoietin) should be avoided within 7 days prior to detection]: Absolute neutrophil count (ANC) ≥1×10^9 /L; hemoglobin ≥70 g/L.; platelets ≥50×10^9 /L; absolute lymphocyte count (ALC) ≥0.3×10^9 /L;
  2. Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×upper limit of normal (ULN); total serum bilirubin ≤ 1.5×ULN.
  3. Kidney function: Serum creatinine ≤2.5×upper limit of normal (ULN), or； Creatinine clearance rate (CrCl) calculated according to Cockcroft-Gault formula ≥ 60 ml/min.
  4. Electrolytes: Serum potassium ≥ 3.0 mmol/L; Serum calcium ≥ 2.0 mmol/L; Serum magnesium ≥ 0.5 mmol/L.
  5. Coagulation function: Fibrinogen ≥ 1.0 g/L; activated partial thromboplastin time (APTT) ≤ ULN+10s, prothrombin time (PT) ≤ ULN+3s.
  6. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%.
* The subjects must be willing to provide valid initial diagnostic evidence and undergo bone marrow examinations before and after treatment.
* Women of childbearing age and all male patients must consent to use a effective contraception for at least 12 months after Meta10-BCMA infusion and until two consecutive PCR tests show no more CAR T cells in vivo；
* The subjects should have measurable disease based on at least one of the following parameters:

  1. The proportion of primitive naive or monoclonal plasma cells ≥ 5% by bone marrow cytology, bone marrow biopsy histology or flow cytometry;
  2. Serum monoclonal protein (M-protein) level: M protein ≥10 g/L for IgG type, M protein ≥5g/L for IgA, IgD, IgM, and IgE type;
  3. Urine M protein level ≥200 mg/24 hours;
  4. Light chain multiple myeloma without measurable lesions in serum or urine: the affected serum free light chain ≥100 mg/L with abnormal serum κ/λ free light chain ratio;
  5. There are measurable extramedullary plasmacytoma lesions.

Exclusion Criteria:

* Treatment with the following therapies within the specified period:

  1. Any hematopoietic stem cell transplant(HSCT) within 2 months prior to the start of infusion of Meta10-BCMA, or any immunosuppressive therapy due to graft-versus-host disease after HSCT within the screening period;
  2. Any major surgery within 4 weeks prior to screening;
  3. Any radiotherapy 2 weeks prior to screening;
  4. Any intrathecal treatment within 1 week prior to the start of infusion of Meta10-BCMA;
  5. Any live vaccination within 4 weeks prior to the start of infusion of Meta10-BCMA and/or plan to receive live vaccines after participation in the trial;
  6. Any clinical trial therapy within 4 weeks prior to the start of infusion of Meta10-BCMA, or ongoing participation in other clinical trials.
* Following disease or surgical history:

  1. ≥ grade 2 arrhythmia according to NCI CTCAE 5.0 grade or QTc> 450 ms (male), QTc> 470ms (female) (QTc is calculated using Fridericia correction formula QTc = QT / RR0.33) subjects with a history of Torsades de pointes ventricular tachycardia or congenital prolonged QT syndrome;
  2. Subjects with any of the following diseases within 12 months before the screening: including but not limited to unstable angina pectoris, myocardial infarction, congestive heart failure and severe arrhythmia, coronary artery bypass grafting or peripheral artery bypass grafting surgery, cerebrovascular events (including transient ischemic attacks), etc.;
  3. Uncontrollable and active infections during the screening period regarded by the investigators;
  4. Subjects infected with human immunodeficiency virus (HIV);
  5. Subjects with active hepatitis B (defined as hepatitis B surface antigen positive or hepatitis B core antibody positive, concomitant hepatitis B virus DNA level > 100 IU/ml);
  6. The hepatitis C virus (HCV) antibody is positive, and the peripheral blood HCV RNA is positive;
  7. Subjects with severe electrolyte disturbance regarded by the investigators;
  8. Subjects with a clear gastrointestinal bleeding tendency, including the following: active local ulcer lesions, and fecal occult blood (≥ ++); subjects with a history of melena and hematemesis within two months prior to screening; Subjects who may have a major gastrointestinal bleeding history;
  9. Subjects with a history of solid organ transplantation;
  10. Subjects with other acute, severe, or chronic medical or psychological conditions regarded by investigators as not suitable for enrollment;
  11. Pregnant or lactating women.
* Prohibited treatment and/or medication:

  1. Ongoing therapy with other anti-tumor drugs, including traditional Chinese medicine;
  2. On-going therapy with drugs that extend the QT interval (including Class Ia and III antiarrhythmic drugs);
  3. Subjects who need to receive oxygen daily;
  4. Long-term use of corticosteroids (except for local inhalation).
* Others:

  1. Subject with a history of psychotropic substance abuse who are unable to quit or have mental disorders;
  2. Subjects with concomitant diseases or comorbidities that could seriously endanger the safety of the patient or affect the completion of the trial as judged by the investigators;
  3. There are not enough unmobilized mononuclear cells available for collection for CAR-T cell production.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
MTD | MTD will be determined based on DLTs observed during the first 35 days of study treatment.
  Determine the Maximal Tolerable Dose(MTD)
Adverse events (AEs) | 1 year post Meta10-BCMA infusion
  Adverse events will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Cmax | 1 year post Meta10-BCMA infusion
  The maximum concentration (Cmax) of CAR-T cell expansion in peripheral blood
Pharmacodynamics | Up to 28 days after infusion
  Concentration levels of CAR-T related serum cytokines such as CRP, IL-6, INF-γ at each time point.
Objective response rate (ORR) | 1 year post Meta10-BCMA infusion
  According to the IMWG 2016 version, evaluate the overall tumor response rate (including sCR, CR, VGPR, PR) and the number of subjects in each dose group and all subjects at 1 month, 3 months, 6 months, 9 months and 12 months after CAR-T treatment.
Overall survival (OS) | 1 year post Meta10-BCMA infusion
  OS is measured from the date of the infusion of Meta10-BCMA to the date of the subjects' death.
Progression-free survival (PFS) | 1 year post Meta10-BCMA infusion
  The time from the start of Meta10-BCMA treatment for the subjects to the first disease progression or death for any reason.
Tmax | 1 year post Meta10-BCMA infusion
  The time to reach the maximum concentration (Tmax)
AUC0-28d | 1 year post Meta10-BCMA infusion
  The area under the curve AUC0-28d at 28 days.
AUC0-90d | 1 year post Meta10-BCMA infusion
  The area under the curve AUC0-90d at 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No